CLINICAL TRIAL: NCT05923320
Title: Effect of an Educational Intervention for Postpartum Mothers on Their Attitudes Towards Childhood Vaccinations and Breastfeeding:
Brief Title: The Effect of Education Given to Postpartum Women on Their Attitudes Towards Childhood Vaccinations and Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AmasyaU18
Record Dates: First submitted 2023-06-07; First posted 2023-06-28 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Breast Feeding; Vaccination Refusal; Training Group, Sensitivity
Keywords: Training; breast-feeding; childhood vaccines; newborn; puerperant woman
MeSH Terms: conditions — Breast Feeding; Vaccination Refusal; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: A repetitive measure design with a pretest-posttest control group
Who Masked: Participant
Masking Description: single paticipant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group -assigned intervention (Experimental): The experimental group was given training on infancy vaccines and breastfeeding. The times of the trainings are determined based on the Postpartum Care Management Guide of the Ministry of Health. In the hospital on the first day after birth, 2-7. days and 30-42. Three days in total, trainings were given on breastfeeding and childhood vaccinations by making home visits. The training content has been prepared by taking into account the Ministry of Health Breastfeeding Guide (5) and the Ministry of Health's vaccination calendar and the Primary Care Vaccine Guide. The trainings will be given to the puerperant women individually. About 30 minutes of training will be given and their questions, if any, will be answered.
  Interventions: Behavioral: training
- control grouup (No Intervention): no training was given to the control group

INTERVENTIONS:
Behavioral: training — The experimental group was given training on infancy vaccines and breastfeeding. The times of the trainings are determined based on the Postpartum Care Management Guide of the Ministry of Health. In the hospital on the first day after birth, 2-7. days and 30-42. Three days in total, trainings were given on breastfeeding and childhood vaccinations by making home visits. The training content has been prepared by taking into account the Ministry of Health Breastfeeding Guide (5) and the Ministry of Health's vaccination calendar and the Primary Care Vaccine Guide. The trainings will be given to the puerperant women individually. About 30 minutes of training will be given and their questions, if any, will be answered.
  Arms: experimental group -assigned intervention

SUMMARY:
Introduction:Breastfeeding and childhood vaccinations are the two most important public health practices for the healthy growth and development of the newborn.

Aim:To investigate the effects of comprehensive training to be given to post-partum women who have just given birth in Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, obstetrics and gynecology service, on their attitudes towards childhood vaccinations and breastfeeding.

Method:This research is in the type of repetitive measurement experimental design with pre-test post-test control group.

The sample consisted of 30 experimental and 30 control groups selected from the universe by computer-assisted randomization method. The experimental group was hospitalized on the first day after birth, on the 2nd-7th day. days and 30-42.

The trainings will be given to the post-partum women individually. About 30 minutes of training will be given and their questions, if any, will be answered. Then, data collection tools will be applied when the babies are 2,4,6 months old (posttest).

Conclusion:This study will enable the comprehensive education to be given to post-partum women who have just given birth in the hospital, to improve their attitudes towards childhood vaccines and to increase the breastfeeding rate.

DETAILED DESCRIPTION:
Introduction:Breastfeeding and childhood vaccinations are the two most important public health practices for the healthy growth and development of the newborn. Although vaccination is one of the most effective and most successful health protection-improvement practices, the cases of vaccine refusal that emerged after 1990 in the world and after 2010 in our country, which increased rapidly, constitute a serious global problem in terms of vaccine-preventable epidemics. is doing. The number of anti-vaccination families has been increasing in recent years. The number of families who do not want to be vaccinated, which was around 1400 in 2014 in our country, is more than 23000 in 2017. If this increase continues like this, it is likely that social immunity will deteriorate and epidemics will occur in the following years. Despite all vaccination campaigns in the world, an average of 1.5 million people die every year from vaccine-preventable diseases.

Aim:To investigate the effects of comprehensive training to be given to post-partum women who have just given birth in Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, obstetrics and gynecology service, on their attitudes towards childhood vaccinations and breastfeeding.

Method:This research is in the type of repetitive measurement experimental design with pre-test post-test control group.

The research will consist of newly delivered post-partum women in Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital gynecology and obstetrics service between 14 March 2022 and September 2023. The universe of the research will consist of all post-partum women who gave birth in the hospital where the research was conducted at the time of the research. The sample consisted of 30 experimental and 30 control groups selected from the universe by computer-assisted randomization method. The experimental group was hospitalized on the first day after birth, on the 2nd-7th day. days and 30-42. Trainings on breastfeeding and childhood vaccinations will be given three times in total by making home visits. The training content has been prepared by taking into account the Ministry of Health Breastfeeding Guide, the Ministry of Health's vaccination schedule, and the Primary Care Vaccination Guide. The trainings will be given to the post-partum women individually. About 30 minutes of training will be given and their questions, if any, will be answered. Then, data collection tools will be applied when the babies are 2,4,6 months old (posttest).

Conclusion:

This study will enable the comprehensive education to be given to post-partum women who have just given birth in the hospital, to improve their attitudes towards childhood vaccines and to increase the breastfeeding rate. It is thought that the results of the study will support the post-partum women, physically, socially and culturally and will guide the programs that will improve the newborns and post-partum women healths.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* 18 and over years old
* Those who volunteered to participate in the study women who do not have communication and mental difficulties

Exclusion Criteria:

* Those who do not fill out the entire questionnaire
* Having a newborn's disease
* Having a postpartum depression

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — puerprant women
Enrollment: 30 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Attitudes of The Evaluation Scale | Change from "Breastfeeding Attitudes of The Evaluation Scale" scores at 6 months
  The highest score that can be obtained from the scale is 184, and as the score from the scale increases, women's attitudes towards breastfeeding are evaluated positively. Sentences with colored (yellow) colors will be scored as "I totally agree" 4-3-2-1-0 as positive attitude, other sentences will be considered negative and reverse scoring will be done as "I totally agree" 0-1-2-3-4. The scale total score is 184. The score of positive items is 88, and the score of negative items is 96. As the score increases, it is evaluated that the breastfeeding attitude is positive.
The Parent Attitudes About childhood vaccines scale (PACV) | Change from "The Parent Attitudes About childhood vaccines scale " scores at 6 months
  It consists of 15 questions. In the first two questions, the participant was asked whether the child was the firstborn and the degree of closeness with the child. The main PACV items start from the 3rd question and consist of a total of 15 items and 3 sub-areas (Question 3-Question 15). These sub-fields are; behavior are general attitudes and safety-efficacy domains. Evaluation scores of the scale; 2 points for hesitant answers, 0 points for unhesitating answers, 1 point for "I'm not sure or I don't know" answers. Items 1 and 2, in which the answer "I don't know" is considered as missing data, are excluded when scoring them, and 2 points are assigned to hesitant responses and 0 points to unhesitating responses for these items. After the scores of each item are given, they are added together;The total raw score is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: duygu murat öztürk, PhD, Principal Investigator — Amasya University
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared